CLINICAL TRIAL: NCT01421888
Title: The NIH UNI Study: Urea Cycle Disorders, Nutrition and Immunity
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110217; 11-HG-0217
Record Dates: First submitted 2011-08-20; First posted 2011-08-23 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2013-04-17

CONDITIONS: Argininosuccinic Aciduria; Carbamoyl-Phosphate Synthase I Deficiency; Citrullinemia; Ornithine Carbamoyltransferase Deficiency; Hyperargininemia; N-Acetylglutamate Synthase Deficiency
Keywords: Immunity; Urea Cycle Disorder; Nutrition; Vaccination; Influenza
MeSH Terms: conditions — Argininosuccinic Aciduria; Citrullinemia; Ornithine Carbamoyltransferase Deficiency Disease; Hyperargininemia; N-acetyl glutamate synthetase deficiency; Urea Cycle Disorders, Inborn; Influenza, Human

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objectives:

* To study nutrition and immune system problems in people with urea cycle disorders.
* To study how people with urea cycle disorders and healthy volunteers respond to standard flu and/or hepatitis A vaccines.
* To compare differences in nutrition and immune systems of people with urea cycle disorders with that of healthy volunteers.

Eligibility:

* Healthy males and females at least 2 years of age who are able to travel to the National Institutes of Health hospital in Bethesda, MD
* Males and females at least 2 years of age who have a urea cycle disorder and are able to travel to the National Institutes of Health hospital in Bethesda, MD.

Design:

For Patients with urea cycle disorder:

* Participants will spend 2 to 3 days in the National Institutes of Health hospital for the following tests:
* A physical exam and review of medical history
* Food log for 3 days before the start of the study
* Blood tests
* 24-hour urine collection
* Resting metabolism test
* DEXA scan imaging study of bones and body fat
* Participants who are old enough to do certain tasks by themselves (like dressing and eating) can choose to have the following extra tests:
* 24-hour metabolic room measurements
* BodPod(Registered Trademark) study to measure bones and body fat
* Participants may choose to have a flu shot and/ or Hepatitis A shot at the end of the study and will be monitored to check for possible side effects.
* Participants will return within 1 to 3 months for follow-up tests/immunizations.

For Healthy Volunteers:

* Participants will be seen at the outpatient clinics at the National Institutes of Health hospital for up to 2 visits for the following:
* Review food log completed 3 days before the start of the study
* Blood tests
* Participants may choose to have a flu shot and/ or Hepatitis A shot at the end of the study and will be monitored to check for possible side effects.
* Participants will return within 1 to 3 months for follow-up tests/immunizations.
* Review of second food log completed 3 days before second outpatient visit

DETAILED DESCRIPTION:
Urea cycle disorders (UCD) are amongst the most frequent of the inborn errors of metabolism (IEM) and result from a block in the hepatic disposal of waste nitrogen from protein catabolism. Viral infections play a significant role in precipitating life-threatening acute hyperammonemic crises in UCD. The recent H1N1 influenza pandemic has placed this vulnerable population at significant risk. The standard of care for these patients is routine vaccination for seasonal and H1N1 influenza viruses. However, nutritional deficiencies and their underlying enzymopathy may affect the efficacy of vaccination.

Dietary management of urea cycle disorders includes dietary modification with protein restriction. Protein energy malnutrition, essential fatty acid deficiencies and micronutrient deficiencies due to restrictive dietary management have been reported in various inborn errors of metabolism. In general, dietary deficiencies and their effect on immune function are well documented.

In addition to the disposal of waste nitrogen, the urea cycle also generates arginine for various biologic functions. Depending on the site of the metabolic block, UCD patients are at risk for becoming systemically deficient in citrulline and arginine, with potential implications for the immune system. The immunomodulatory roles of the amino acids citrulline and arginine have been characterized in the context of nutritional deficiencies in disease states such as cancer and sepsis. Systemic infection may also deplete systemic citrulline and arginine, compounding an underlying deficiency in UCD. Cells of the immune system have a more direct relationship with the urea cycle: urea cycle enzymes arginosuccinate synthetase (ASS), arginosuccinate lyase (ASL) and arginase (ARG1) may also be components of leukocyte metabolism. Overall, general and specific nutritional deficiencies and enzymopathies affecting leukocyte metabolism may potentially affect vaccine efficacy. However, immune system function in experiments of nature such as UCD remains an understudied area.

In this protocol, we will clinically evaluate the nutritional/metabolic and immunologic states of patients with UCD or related disorders. Routine inpatient admissions will last 2-3 days and involve urine collection, blood drawing, radiological procedures, nutrition assessment and biometrics, and vaccination for combined seasonal/H1N1 influenza. Follow-up outpatient appointments will be scheduled at the end of the study period.

The study objectives will be to describe the nutritional and immune deficiencies seen, query for nutrition/enzymatic/immunologic correlations in this patient population, describe vaccine efficacy in this patient population, and search for new genes in rare families that have evidence for an unknown class of UCD. The population will consist of patients previously evaluated at NIH, physician referrals, and families directed to the study from clinicaltrials.gov as well as the National Urea Cycle Disorders Foundation. All patients will be evaluated at the NIH Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

Any gender and ethnicity age 2 years and older with a diagnosis of a urea cycle disorder are eligible to enroll in this protocol.

Patients need to be medically and nutritionally managed by a local metabolic provider. If necessary, we will obtain written consent from the patient to review medical records from their home physician to confirm eligibility.

Healthy Volunteers:

Any gender and ethnicity age 2 years and older are eligible to enroll in this protocol.

Have access to own personal medical provider <TAB>

EXCLUSION CRITERIA:

Less than 2 years of age

Inability to travel to NIH because of their medical condition

Recent (6 month) history of vaccination or immune modulating drug

Severe reactions to eggs and or latex

History of severe reactions to previous immunizations (e.g. hives, rash, difficulty breathing)

Persons without a personal medical provider

Persons with current infections or under care of medical provider for an ongoing medical issue

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-08-08; Study Completion 2013-04-17

CONTACTS AND LOCATIONS:
Overall Officials: Peter J McGuire, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barshop BA, Summar ML. Attitudes regarding vaccination among practitioners of clinical biochemical genetics. Mol Genet Metab. 2008 Sep-Oct;95(1-2):1-2. doi: 10.1016/j.ymgme.2008.08.001. No abstract available. PMID 18816884
- [Background] Batshaw ML, Brusilow S, Waber L, Blom W, Brubakk AM, Burton BK, Cann HM, Kerr D, Mamunes P, Matalon R, Myerberg D, Schafer IA. Treatment of inborn errors of urea synthesis: activation of alternative pathways of waste nitrogen synthesis and excretion. N Engl J Med. 1982 Jun 10;306(23):1387-92. doi: 10.1056/NEJM198206103062303. PMID 7078580
- [Background] Summar M, Tuchman M. Proceedings of a consensus conference for the management of patients with urea cycle disorders. J Pediatr. 2001 Jan;138(1 Suppl):S6-10. doi: 10.1067/mpd.2001.111831. PMID 11148544